CLINICAL TRIAL: NCT06860646
Title: Hospital Registry of Patients with Myocardial Infarction in Individuals Aged 75 Years and Older
Brief Title: Myocardial Infarction in the Elderly
Status: Recruiting | Type: Observational
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 0922142025
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Infarction (MI)
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
An observational registry study of patients aged 75 years and older with an established diagnosis of myocardial infarction, initiated in 2020, with an assessment of clinical, instrumental, demographic and prognostic data. Statistical analysis was performed using the StatTech v. 4.5.0 program (developer - StatTech LLC, Russia). Differences were considered statistically significant at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

- age 75 years and older, presence of an established diagnosis of myocardial infarction at the time of hospitalization.

Exclusion Criteria:

-

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients hospitalized in the State Budgetary Institution of the Ryazan Region "Regional Clinical Cardiology Dispensary" with an established diagnosis of myocardial infarction
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
all-cause death, myocardial infarction, stroke, unplanned percutaneous coronary | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- State Budgetary Institution of the Ryazan Region "Regional Clinical Cardiology Dispensary", Ryazan, Russia

IPD SHARING:
Plan to Share IPD: No